CLINICAL TRIAL: NCT06646887
Title: Comparison of Different Electroporation Systems in the Ablation Treatment of Atrial Fibrillation
Acronym: PFA Champion
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Ana Jordan, Principal Investigator, University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dubrava; 2024/0828-4 (Other: UHDubrava)
Record Dates: First submitted 2024-10-02; First posted 2024-10-17 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-01

CONDITIONS: AF; Ablation of Atrial Fibrillation
MeSH Terms: interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Varipluse, (Active Comparator): Varipulse Arm - Participants in this arm will undergo ablation using the Varipulse system
  Interventions: Other: Electroporation
- PulseSelect (Active Comparator): PulseSelect Arm - Participants in this arm will receive treatment with the PulseSelect system
  Interventions: Other: Electroporation
- Farpulse (Active Comparator): Farapulse Arm - Participants in this arm will undergo ablation using the Farapulse electroporation system.
  .
  Interventions: Other: Electroporation

INTERVENTIONS:
Other: Electroporation — Unlike traditional thermal ablation techniques such as radiofrequency (RF) and cryoablation, the electroporation systems used in this study rely on pulsed electric fields (PEF) to selectively target and ablate cardiac tissue. This non-thermal mechanism reduces the risk of collateral damage to nearby structures, such as the esophagus, phrenic nerve, and coronary arteries.

SUMMARY:
The participant is invited to participate in a clinical study comparing three different techniques for treating atrial fibrillation (AF) called electroporation systems. Atrial fibrillation is an irregular heartbeat that can cause complications if left untreated. The goal of this study is to determine which electroporation system is the most effective and safest for treating AF. These systems work by using electrical energy to disrupt abnormal heart tissue, helping to restore a normal heart rhythm.

DETAILED DESCRIPTION:
The investigators are testing three different electroporation systems: Farapulse, PulseSelect, and Varipulse. Each of these systems uses a similar approach to treat AF, but they may work slightly differently. The investigators want to find out which one is best at permanently stopping the irregular heart rhythm, while also being the safest for patients.

What will happen during the study?

The patient will have two procedures:

First procedure: This is the initial ablation, where the doctors will use one of the three electroporation systems to treat the atrial fibrillation. During this procedure, the investigators will map the heart using a special tool to see exactly where the irregular rhythm is happening.

Second procedure: After about 3 months, the participant will return for a re-mapping procedure. This will allow the doctors to check if the treatment was successful and if any abnormal rhythms have come back. If necessary, the investigator will perform another ablation to correct any remaining problems.

Is it safe? All procedures are performed by experienced doctors who specialize in treating AF. Like any medical procedure, there are some risks, such as small chances of blood clots, injury to nearby tissues, or complications from the anesthesia. However, the electroporation systems are designed to minimize these risks, and the study will closely monitor your loved one for any complications.

What are the benefits of participating? The participant could benefit from receiving one of the latest treatments for atrial fibrillation. By participating, they will help doctors learn which system works best, which could help future patients with similar conditions. Additionally, the participant heart rhythm will be closely monitored, and if any problems arise, they will receive immediate care.

How long will it take? The study will last about 6 to 7 months, with the initial procedure taking place in the next few weeks and a follow-up re-mapping procedure approximately 12-14 weeks later.

ELIGIBILITY:
Patients with symptomatic paroxysmal or persistent atrial fibrillation. Eligible for catheter ablation as per current guidelines. Willing to undergo both an initial ablation procedure and a repeat mapping/ablation if required.

Exclusion Criteria:

Patients with prior ablation procedures. Contraindications for AF ablation (e.g., severe coagulopathy, left atrial appendage thrombus).

Significant comorbidities impacting study outcomes.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness and durability of the ablation procedure. | Three months
  The percentage of patients who achieve complete and durable pulmonary vein isolation without reconnection, confirmed during the re-mapping procedure performed approximately 12-14 weeks after the initial ablation.

CONTACTS AND LOCATIONS:
Locations (2):
- Croatia (2):
  - Clinical Hospital Dubrava, Department of Cardiology, Zagreb, City of Zagreb
  - UHDubrava, Zagreb

IPD SHARING:
Plan to Share IPD: No
Patient Privacy and Confidentiality: Sharing detailed individual data can raise concerns about the privacy of participants. Even with de-identification, there may be a risk of re-identifying participants, especially with a relatively small sample size and specific medical conditions like atrial fibrillation.
  Ethical Considerations: Ethical guidelines often require that participant data is protected and only used for the specific purposes outlined in the consent forms. Sharing IPD might exceed the scope of what participants agreed to when they enrolled in the study.
  Regulatory Restrictions: Some regulatory bodies or institutions may impose strict guidelines on the sharing of sensitive medical data to prevent misuse or ensure data security, particularly when dealing with experimental procedures or novel technologies like electroporation systems.

REFERENCES:
- [Background] Reddy VY, Dukkipati SR, Neuzil P, Anic A, Petru J, Funasako M, Cochet H, Minami K, Breskovic T, Sikiric I, Sediva L, Chovanec M, Koruth J, Jais P. Pulsed Field Ablation of Paroxysmal Atrial Fibrillation: 1-Year Outcomes of IMPULSE, PEFCAT, and PEFCAT II. JACC Clin Electrophysiol. 2021 May;7(5):614-627. doi: 10.1016/j.jacep.2021.02.014. Epub 2021 Apr 28. PMID 33933412